CLINICAL TRIAL: NCT05524402
Title: Live Video Mind-body Treatment to Prevent Persistent Symptoms Following mTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jonathan Greenberg, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022P001521; K23AT010653-01A1 (NIH)
Record Dates: First submitted 2022-08-17; First posted 2022-09-01 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: MTBI - Mild Traumatic Brain Injury; Anxiety
Keywords: MTBI - Mild Traumatic Brain Injury; Anxiety; Mindfulness
MeSH Terms: conditions — Brain Concussion; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOR-C 1 (Experimental): TOR-C 1 is an active intervention adapted from the original Toolkit for Optimal Recovery program, adjusted for patients with mTBI and anxiety. The TOR-C 1 sessions address mind-body skills, including eliciting the relaxation response (eg, body scan, deep breathing, mindfulness), cognitive-behavioral strategies (eg, reframing), acceptance and commitment skills (eg, acceptance), and skills for returning to activity (eg, goal setting, activity pacing). The format is a 4-week program delivered over live video with weekly sessions and home practice.
  Interventions: Behavioral: TOR-C 1
- TOR-C 2 (Active Comparator): TOR-C 2 is an active intervention teaching educational information on key modifiable factors relating to recovery after concussion, such as return to activity, the role of nutrition and sleep, and the relationship between concussion and anxiety. The format is a 4-week program delivered over live video with weekly sessions.
  Interventions: Behavioral: TOR-C 2

INTERVENTIONS:
Behavioral: TOR-C 1 — TOR-C 1 is an active intervention, adapted from the original Toolkit for Optimal Recovery program, adjusted for patients with mTBI and anxiety. The TOR-C 1 sessions address mind-body skills, including eliciting the relaxation response (eg, body scan, deep breathing, mindfulness), cognitive-behavioral strategies (eg, reframing), acceptance and commitment skills (eg, acceptance), and skills for returning to activity (eg, goal setting, activity pacing). The format is a 4-week program with weekly sessions and home practice.
  Arms: TOR-C 1
Behavioral: TOR-C 2 — TOR-C 2 is an active intervention teaching educational information on key modifiable factors relating to recovery after concussion, such as return to activity, the role of nutrition and sleep, and the relationship between concussion and anxiety. The format is a 4-week program delivered over live video with weekly sessions.
  Arms: TOR-C 2

SUMMARY:
The investigator aims to conduct a pilot randomized controlled trial to test the feasibility of two symptom management programs for college-age individuals with recent concussions and anxiety, TOR-C 1 and TOR-C 2. The investigator will assess the feasibility of recruitment procedures (screening, eligibility, and enrollment) and data collection as well as the feasibility, credibility, and acceptability of the programs (adherence, retention, fidelity, and satisfaction), following prespecified benchmarks. Both programs will be delivered virtually (Zoom).

DETAILED DESCRIPTION:
The investigator aims to conduct a pilot randomized controlled trial to test the feasibility of two symptom management programs for college-age individuals with recent concussions and anxiety, TOR-C 1 and TOR-C 2. The investigator will assess the feasibility of recruitment procedures (screening, eligibility, and enrollment) and data collection as well as the feasibility, credibility, and acceptability of the programs (adherence, retention, fidelity, and satisfaction), following prespecified benchmarks. Both programs will be delivered virtually (Zoom).

Each program will consist of four 45-minute sessions over the secure Zoom platform. Participants will receive a treatment manual. There are 3 assessment points consisting of self-report surveys: baseline, post program, and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, ages 18-35
* English fluency and literacy
* Diagnosed with a concussion in the past 10 weeks
* Owns a smartphone or computer with Internet access
* Willingness and ability to participate in four 45-minute program sessions and answer remote questionnaires before, after, and 3-month following the program
* Free of concurrent psychotropic or have been on stable dosage for at least 6 weeks
* Clinically significant anxiety symptoms (score ≥ 5 on GAD-7 anxiety scale)

Exclusion Criteria:

* Previous history of moderate or severe TBI OR concussion in the past 2 years that resulted in symptoms lasting 3 months or more
* Diagnosed with a medical illness expected to worsen in the next 6 months (e.g., malignancy)
* Lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder
* Current substance abuse or dependence and current substance use disorder
* Current active self-reported suicidal ideation
* Practice of mindfulness techniques for greater than 45 minutes per week within the last 3 months
* Participation in a mind-body or CBT treatment in the past 3 months
* Currently pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Greenberg, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenberg J, Singh T, Iverson GL, Silverberg ND, Macklin EA, Parker RA, Giacino JT, Yeh GY, Vranceanu AM. A Live Video Mind-Body Treatment to Prevent Persistent Symptoms Following Mild Traumatic Brain Injury: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2021 Jan 14;10(1):e25746. doi: 10.2196/25746. PMID 33443484
- [Derived] Greenberg J, Levey NS, Becker M, Yeh GY, Giacino JT, Iverson G, Silverberg ND, Parker RA, Vranceanu AM. Feasibility Randomized Controlled Trial of the Toolkit for Optimal Recovery After Concussion: A Live Video Program to Prevent Persistent Concussion Symptoms in Young Adults With Anxiety. Arch Phys Med Rehabil. 2025 Apr;106(4):527-536. doi: 10.1016/j.apmr.2024.10.011. Epub 2024 Nov 5. PMID 39505248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited via provider and self-referrals from the MGH Sports Concussion Clinic and Emergency Department, as well as concussion clinics nationwide, college health resources (e.g., sports medicine centers), relevant public social media sites (e.g., Facebook), Research Invitations via Patient Gateway after identifying potential participants through Research Patient Database Registry (RPDR) queries, and MGB Rally.
Pre-assignment Details: Of the 51 eligible patients, 50 enrolled and were randomized.
Period: Overall Study
Arm/Group | TOR-C 1 | TOR-C 2
Started | 25 | 25
Post-Test (4 Weeks) | 22 | 24
Follow-Up (12 Weeks) | 20 | 23
Completed | 20 | 23
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is same as indicated in "Participant Flow".
Groups:
- Total: Total of all reporting groups
Arm/Group | TOR-C 1 | TOR-C 2 | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.64 (4.83) | 23.28 (4.56) | 23.45 (4.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 23 | 19 | 42
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 21 | 21 | 42
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50
Numerical Rating Scale - During Activity [Mean (Standard Deviation); unit: units on a scale] — Rate of pain during activity using a Likert scale with 0 being no pain and 10 being worst possible pain.
  units on a scale | 4.12 (2.91) | 5.20 (2.24) | 4.66 (2.62)
Post-Concussion Symptom Scale [Mean (Standard Deviation); unit: units on a scale] — Rate post-concussion symptoms on a 1 to 6-point Likert scale. Total scores range from 22 to 132, with higher scores indicating worse concussion symptoms.
  units on a scale | 43.52 (31.26) | 50.61 (23.92) | 46.99 (27.85)
Generalized Anxiety Disorder Scale (GAD-7) [Mean (Standard Deviation); unit: units on a scale] — 7-item questionnaire measuring symptoms of anxiety within the past 2 weeks on a scale of 0 to 3. Total scores range from 0 to 21 and higher scores indicate more symptoms of anxiety.
  units on a scale | 10.00 (4.85) | 13.48 (4.57) | 11.74 (4.98)
Hospital Anxiety And Depression Scale (HADS) - Anxiety Subscale [Mean (Standard Deviation); unit: units on a scale] — 7-item anxiety subscale of the Hospital Anxiety and Depression Scale. Scores range from 0-21, with higher scores indicating more symptoms. Scores greater than 8 indicate clinically significant symptoms.
  units on a scale | 9.46 (3.63) | 11.80 (4.05) | 10.63 (3.99)
World Health Organization - Disability Assessment Schedule 2.0 (WHODAS) [Mean (Standard Deviation); unit: units on a scale] — The WHODAS 2.0 measures level of functioning in six domains: cognition, mobility, self-care, getting along, life activities, and participation. Each item is on the scale is measured 0-4, with total scores ranging from 0 to 48. Higher scores indicate more disability (worse outcomes).
  units on a scale | 13.47 (9.96) | 16.29 (8.80) | 14.88 (9.41)
Fear Avoidance Behavior After Traumatic Brain Injury (FAB-TBI) [Mean (Standard Deviation); unit: units on a scale] — A 16-item questionnaire assessing beliefs about how work and physical activities affect mTBI symptoms, and whether they should be avoided on a scale of 0 to 3. Total scores range from 0 to 48 and higher scores represent higher fear avoidance.
  units on a scale | 39.01 (11.50) | 44.45 (9.46) | 41.80 (10.76)
Pain Catastrophizing Scale (PCS) [Mean (Standard Deviation); unit: units on a scale] — A 13-item questionnaire assessing one's tendency to focus on pain-related thoughts and feel helpless and hopeless due to pain on a scale of 0 to 4. Total scores range from 0 to 25 and higher scores indicate higher pain catastrophizing (worse outcomes).
  units on a scale | 17.13 (14.26) | 20.64 (14.78) | 18.92 (14.48)
Cognitive And Affective Mindfulness Scale-Revised (CAMS-R) [Mean (Standard Deviation); unit: units on a scale] — Measures participant's broad conceptualization of mindfulness, items range from 1-4 and total scores range from 12-48, with higher values reflecting higher levels of mindfulness
  units on a scale | 29.31 (5.39) | 27.24 (5.05) | 28.28 (5.28)
Behavioral Response To Illness (BRIQ) - All-or-Nothing Subscale [Mean (Standard Deviation); unit: units on a scale] — A 6-item subscale of the BRIQ measuring "all or nothing behaviors" (tendency for overexertion). This subscale is rated on a scale of 0 to 4, with higher scores indicating more all or nothing behavior. Total scores on this subscale range from 0 to 24.
  units on a scale | 11.64 (5.30) | 12.84 (5.24) | 12.24 (5.25)
Hospital Anxiety And Depression Scale (HADS) - Depression Subscale [Mean (Standard Deviation); unit: units on a scale] — 7-item depression subscale of the Hospital Anxiety and Depression Scale. Scores range from 0-21, with higher scores indicating more symptoms. Scores greater than 8 indicate clinically significant symptoms.
  units on a scale | 6.02 (4.68) | 8.22 (4.02) | 7.12 (4.46)
Behavioral Response To Illness (BRIQ) - Limiting Behaviors Subscale [Mean (Standard Deviation); unit: units on a scale] — A 7-item subscale of the BRIQ measuring "limiting behaviors" (frequency of inactivity). This subscale is rated on a scale of 0 to 4, with total scores ranging from 0 to 28. Higher scores indicate more limiting behavior (worse outcomes).
  units on a scale | 14.88 (7.22) | 17.28 (4.98) | 16.08 (6.26)
Numerical Rating Scale - At Rest [Mean (Standard Deviation); unit: units on a scale] — Participant's pain at rest using a Likert scale with 0 being no pain and 10 being worst possible pain. Higher scores indicate worse pain severity.
  units on a scale | 3.20 (2.50) | 3.72 (2.26) | 3.46 (2.35)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Scored Above the Midpoint on Each Subscale of the Credibility and Expectancy Questionnaire (CEQ)
Description: Assessed using the Credibility and Expectancy Questionnaire (CEQ) which asks the participant indicate how much they believe, right now, that the intervention they will receive will help manage their concussion and related worry. Possible scores on both the credibility and expectancy subscales range from 3 to 27 and have a midpoint score of 14. The number of participants that scored at or above 14 on the credibility and/or expectancy subscales are reported below.
Time Frame: Baseline (0 Weeks)
Population: The total of participants (separated by condition) that scored above the midline on the credibility and expectancy subscales of the Credibility and Expectancy Questionnaire (CEQ).
Measure: Count of Participants; unit: Participants
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
Participants
  Credibility Subscale | 21 | 23
  Expectancy Subscale | 16 | 19

2. Primary Outcome: Number of Participants Who Scored Above the Midpoint on the Client Satisfaction Scale
Description: Measured using the Client Satisfaction Scale which assess participants' satisfaction with participation in the study. The score range is 0-12. Higher scores indicate greater satisfaction.
Time Frame: Post-Test (4 Weeks)
Population: The proportion of participants that completed the post-test and scored above the midpoint on the Client Satisfaction Scale.
Measure: Count of Participants; unit: Participants
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 21 | 23
Participants | 20 | 20

3. Primary Outcome: Feasibility of Recruitment
Description: Rate at which recruitment was possible
Time Frame: Baseline (0 Weeks)
Population: The proportion of eligible patients (n=54) who agree to participate (n=50).
Measure: Count of Participants; unit: Participants
Groups:
- Total: Outcome calculated for entire sample (TOR-C1 and TOR-C2; n=50).
Arm/Group | Total
Number analyzed (Participants) | 54
Participants | 50

4. Primary Outcome: Acceptability of Treatment
Description: Rate at which program was accepted, measured by attendance.
Time Frame: Post-Test (4 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
Participants | 21 | 23

5. Primary Outcome: Adherence to Homework
Description: Rate of participant's completion of homework assigned (practicing at least 1 program skill, 3 days/week on average) throughout the study.
Time Frame: Collected during intervention, an average of 4 weeks
Population: Sample represents the number of TOR-C1 program completers (i.e., those who attended at least 3 of 4 program sessions).
Measure: Count of Participants; unit: Participants
Groups:
- TOR-C1: TOR-C 1 is an active intervention adapted from the original Toolkit for Optimal Recovery program, adjusted for patients with mTBI and anxiety. The TOR-C 1 sessions address mind-body skills, including eliciting the relaxation response (eg, body scan, deep breathing, mindfulness), cognitive-behavioral strategies (eg, reframing), acceptance and commitment skills (eg, acceptance), and skills for returning to activity (eg, goal setting, activity pacing). The format is a 4-week program delivered over live video with weekly sessions and home practice.
Arm/Group | TOR-C1
Number analyzed (Participants) | 21
Participants | 16

6. Primary Outcome: Therapist Adherence
Description: Rate of interventionist's delivering the programs by following the established session topics and practices
Time Frame: Collected during intervention, an average of 4 weeks
Population: 20% (n=10) of session recordings for each condition were randomly selected for clinician fidelity checks. The clinician is evaluated on the degree to which they delivered session content as intended with adequate clinical skills. Each subcomponent in each session is scored on a 1-5 point scale. The overall average score for the randomly selected TOR-C1 and TOR-C2 sessions is then assessed to produce an average percent of therapist adherence for each intervention.
Measure: Mean (Standard Deviation); unit: percentage of adherence
Units Other Than Participants: Program Sessions
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
Number analyzed (Program Sessions) | 10 | 10
percentage of adherence | 96.30 (0.60) | 97.60 (0.43)

7. Primary Outcome: Feasibility of Assessments at Baseline
Description: Rate of participant's completion of self-report measures, with no measures missing
Time Frame: Baseline (0 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
Participants | 25 | 25

8. Primary Outcome: Feasibility of Assessments at Post-Test
Description: Rate of participant's completion of self-report measures, with no measures missing
Time Frame: Post-Test (4 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
Participants | 22 | 24

9. Primary Outcome: Feasibility of Assessments at Follow-up
Description: Rate of participant's completion of self-report measures, with no measures missing
Time Frame: Follow-up (12 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
Participants | 20 | 23

10. Primary Outcome: Adverse Events
Description: Any self reported or observed negative events related to participation
Time Frame: Collected during intervention, an average of 4 weeks
Measure: Number; unit: Adverse events related to participation
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
Adverse events related to participation | 0 | 0

11. Secondary Outcome: Numerical Rating Scale
Description: Rate of a participant's pain at rest and with activity using a Likert scale with 0 being no pain and 10 being worst possible pain.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-Up (12 Weeks)
Population: Analysis population consists of measure completers (subject to change at each assessment point)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline - During activity | 4.12 (2.91) | 5.20 (2.24)
  Baseline - At rest | 3.20 (2.50) | 3.72 (2.26)
  Post-Test - During activity: number analyzed (Participants) | 22 | 24
  Post-Test - During activity | 1.91 (1.57) | 3.50 (2.27)
  Post-Test - At rest: number analyzed (Participants) | 22 | 24
  Post-Test - At rest | 1.45 (1.30) | 2.38 (1.74)
  Follow-Up - During activity: number analyzed (Participants) | 20 | 23
  Follow-Up - During activity | 1.40 (2.01) | 2.35 (2.10)
  Follow-Up - At rest: number analyzed (Participants) | 20 | 23
  Follow-Up - At rest | 1.15 (1.46) | 1.43 (1.24)

12. Secondary Outcome: Post-Concussion Symptom Scale (PCSS)
Description: The PCSS measures post-concussion symptoms on a 1-6-point Linkert scale. Higher scores represent greater symptom severity and total scores can range from 22 to132 points.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-Up (12 Weeks)
Population: Analysis population consists of measure completers (subject to change at each assessment point)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 43.52 (31.26) | 50.61 (23.92)
  Post-Test: number analyzed (Participants) | 22 | 24
  Post-Test | 12.50 (7.57) | 29.08 (24.05)
  Follow-Up: number analyzed (Participants) | 20 | 23
  Follow-Up | 11.65 (11.26) | 23.13 (24.12)

13. Secondary Outcome: Generalized Anxiety Disorder Scale (GAD-7)
Description: 7-item questionnaire measuring symptoms of anxiety within the past 2 weeks on a scale of 0 to 3. Total scores range from 0 to 21 and higher scores indicate more symptoms of anxiety.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-Up (12 Weeks)
Population: Analysis population consists of measure completers (subject to change at each assessment point)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 10.00 (4.85) | 13.48 (4.57)
  Post-Test: number analyzed (Participants) | 22 | 24
  Post-Test | 5.00 (3.82) | 7.92 (5.27)
  Follow-Up: number analyzed (Participants) | 20 | 23
  Follow-Up | 3.85 (3.70) | 6.74 (6.45)

14. Secondary Outcome: Hospital Anxiety And Depression Scale (HADS)
Description: Measures symptoms of emotional distress and estimates diagnoses. The scale has 14 items, 7 assess anxiety and 7 depression. Scores range from 0-21 on each subscale, wtih higher scores indicating more symptoms. Scores greater than 8 indicate clinically significant symptoms.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-Up (12 Weeks)
Population: Analysis population consists of measure completers (subject to change at each assessment point)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline - Anxiety | 9.46 (3.63) | 11.80 (4.05)
  Baseline - Depression | 6.02 (4.68) | 8.22 (4.02)
  Post-Test - Anxiety: number analyzed (Participants) | 22 | 24
  Post-Test - Anxiety | 7.81 (4.22) | 8.79 (4.35)
  Post-Test - Depression: number analyzed (Participants) | 22 | 24
  Post-Test - Depression | 3.73 (3.63) | 5.13 (2.63)
  Follow-Up - Anxiety: number analyzed (Participants) | 20 | 23
  Follow-Up - Anxiety | 6.80 (3.97) | 8.39 (5.22)
  Follow-Up - Depression: number analyzed (Participants) | 20 | 23
  Follow-Up - Depression | 2.10 (2.59) | 5.12 (2.96)

15. Secondary Outcome: World Health Organization - Disability Assessment Schedule 2.0 (WHODAS)
Description: The WHODAS 2.0 measures level of functioning in six domains: cognition, mobility, self-care, getting along, life activities, and participation. Each item is on the scale is measured 0-4, with total scores ranging from 0 to 48. Higher scores indicate more disability (worse outcomes).
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-Up (12 Weeks)
Population: Analysis population consists of measure completers (subject to change at each assessment point)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 13.47 (9.96) | 16.29 (8.80)
  Post-Test: number analyzed (Participants) | 22 | 24
  Post-Test | 5.61 (6.32) | 9.83 (8.30)
  Follow-Up: number analyzed (Participants) | 20 | 23
  Follow-Up | 3.10 (3.01) | 7.61 (8.60)

16. Secondary Outcome: Fear Avoidance Behavior After Traumatic Brain Injury (FAB-TBI)
Description: A 16-item questionnaire assessing beliefs about how work and physical activities affect mTBI symptoms, and whether they should be avoided on a scale of 0 to 3. Total scores range from 0 to 48 and higher scores represent higher fear avoidance.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-Up (12 Weeks)
Population: Analysis population consists of measure completers (subject to change at each assessment point)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 24 | 25
score on a scale
  Baseline | 39.01 (11.50) | 44.45 (9.46)
  Post-Test: number analyzed (Participants) | 22 | 24
  Post-Test | 24.51 (7.78) | 36.02 (12.02)
  Follow-Up: number analyzed (Participants) | 20 | 23
  Follow-Up | 24.20 (9.80) | 31.35 (12.19)

17. Secondary Outcome: Pain Catastophizing Scale (PCS)
Description: A 13-item questionnaire assessing one's tendency to focus on pain-related thoughts and feel helpless and hopeless due to pain on a scale of 0 to 4. Total scores range from 0 to 25 and higher scores indicate higher pain catastrophizing (worse outcomes).
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-Up (12 Weeks)
Population: Analysis population consists of measure completers (subject to change at each assessment point)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 17.13 (14.26) | 20.64 (14.78)
  Pose-Test: number analyzed (Participants) | 22 | 24
  Pose-Test | 8.44 (9.37) | 14.46 (13.41)
  Follow-Up: number analyzed (Participants) | 20 | 23
  Follow-Up | 7.80 (9.57) | 13.22 (5.82)

18. Secondary Outcome: Cognitive And Affective Mindfulness Scale-Revised (CAMS-R)
Description: Rate of a participant's broad conceptualization of mindfulness, items range from 1-4 and scores range from 12-48, with higher values reflecting higher levels of mindfulness
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-Up (12 Weeks)
Population: Analysis population consists of measure completers (subject to change at each assessment point)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 29.31 (5.39) | 27.24 (5.05)
  Post-Test: number analyzed (Participants) | 22 | 24
  Post-Test | 33.68 (6.71) | 30.21 (6.74)
  Follow-Up: number analyzed (Participants) | 20 | 23
  Follow-Up | 33.65 (4.80) | 31.13 (5.82)

19. Secondary Outcome: Behavioral Response To Illness (BRIQ) - Limiting Behaviors Subscale
Description: A 7-item subscale of the BRIQ measuring "limiting behaviors" (frequency of inactivity). This subscale is rated on a scale of 0 to 4, with total scores ranging from 0 to 28. Higher scores indicate more limiting behavior (worse outcomes).
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-Up (12 Weeks)
Population: Analysis population consists of measure completers (subject to change at each assessment point)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 14.88 (7.22) | 17.28 (4.98)
  Post-Test: number analyzed (Participants) | 22 | 24
  Post-Test | 6.14 (5.58) | 11.00 (6.41)
  Follow-Up: number analyzed (Participants) | 20 | 23
  Follow-Up | 4.99 (4.30) | 9.83 (7.21)

20. Secondary Outcome: Behavioral Response To Illness (BRIQ) - All-or-Nothing Subscale
Description: A 6-item subscale of the BRIQ measuring "all or nothing behaviors" (tendency for overexertion). This subscale is rated on a scale of 0 to 4, with higher scores indicating more all or nothing behavior. Total scores on this subscale range from 0 to 24.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-Up (12 Weeks)
Population: Analysis population consists of measure completers (subject to change at each assessment point)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TOR-C 1 | TOR-C 2
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline | 11.64 (5.30) | 12.84 (5.24)
  Post-Test: number analyzed (Participants) | 22 | 24
  Post-Test | 8.19 (5.79) | 10.79 (4.90)
  Follow-Up: number analyzed (Participants) | 19 | 23
  Follow-Up | 7.16 (4.95) | 9.52 (6.81)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment (0 weeks) through the follow-up assessment (3 months)
Description: Adverse Event Monitoring: Throughout the study, subjects were monitored for the occurrence of adverse/other events. Lack of effect of treatment is not considered an event. All adverse events will be reported on an adverse event form. The Principle Investigator had the responsibility of reporting serious adverse events (death, life-threatening illness or injury, serious injury, or permanent disability) to PHRC within 24-72 hours of notification.
Arm/Group | TOR-C 1 | TOR-C 2
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT05524402/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT05524402/SAP_001.pdf
  • Informed Consent Form (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT05524402/ICF_002.pdf